CLINICAL TRIAL: NCT00667719
Title: A 28 to 54-week, Open-label, Multicenter Study to Assess the Long-term Safety and Tolerability of the Combination of Aliskiren / Amlodipine / Hydrochlorothiazide in Patients With Essential Hypertension
Brief Title: A Long Term Safety Study to Test the Combination of Aliskiren/ Amlodipine / Hydrochlorothiazide in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSAH100A2301; 2008-001242-10 (EudraCT Number)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; High blood pressure
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — aliskiren; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aliskiren/Amlodipine/Hydrochlorothiazide (Experimental): Participants received aliskiren 300 milligrams (mg) plus hydrochlorothiazide 12.5 mg for one week, at Week 1 followed by combination of aliskiren 300 mg plus amlodipine 5 mg plus hydrochlorothiazide 12.5 mg for one week, at Week 2. Following Week 2, participants were force titrated up to aliskiren 300 mg plus amlodipine 10 mg plus hydrochlorothiazide 25 mg for 26 to 52 weeks (Weeks 28 to 54). All study medications were taken orally with water, once daily in the morning.
  Interventions: Drug: Aliskiren; Drug: Amlodipine; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Aliskiren — 300 mg tablet
Drug: Amlodipine — 5 mg tablet
Drug: Hydrochlorothiazide — 12.5 mg and 25 mg capsule

SUMMARY:
This study tested the safety of the combination of aliskiren/amlodipine/hydrochlorothiazide in participants with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 years of age or older
* Male or female participants are eligible.
* Mean sitting diastolic blood pressure (msDBP) and mean sitting systolic blood pressure (msSBP) Requirements:

  * For newly diagnosed/untreated participants, msDBP ≥ 100 and < 120 millimeters of mercury (mmHg), and/or msSBP ≥ 160 and < 200 mmHg at Visit 1 and Visit 2.
  * For previously treated participants, msDBP ≥ 100 and < 120 mmHg, and/or msSBP ≥ 160 and < 200 mmHg at Visit 2, Visit 3, or Visit 4.
* For participants requiring tapering off their previous antihypertensive medication, they must meet the above criteria and completely discontinue all antihypertensive treatment prior to entering the treatment phase of the study.
* Participants who are eligible and able to participate in the study, and who consent to do so after the purpose and nature of the investigation has been clearly explained to them (written informed consent).

Exclusion Criteria:

* Inability to discontinue all prior antihypertensive medications safely for a period of 1 week to 4 weeks as required by the protocol.
* Participants on three antihypertensive drugs with msDBP ≥ 110 mmHg and/or msSBP ≥ 180 mmHg at Visit 1.
* Participants on four or more antihypertensive drugs at Visit 1.
* Participants with an msSBP ≥ 200 and msDBP ≥ 120 mmHg anytime during the washout period of the study Visit 1-4 must be discontinued from the study.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (>= 5 milli-international units per milliliter mIU/mL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2008-06-05 (Actual); Primary Completion 2009-10-05 (Actual); Study Completion 2009-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (8):
- Investigative Site, Houston, Texas, United States
- Investigative Site, Belgium, Belgium
- Investigative Site, Egypt, Egypt
- Investigative Site, Germany, Germany
- Investigative Site, Poland, Poland
- Investigative Site, Slovakia, Slovakia
- Investigative Site, Spain, Spain
- Investigative Site, Turkey, Turkey (Türkiye)

REFERENCES:
- [Result] Murray AV, Koenig W, Garcia-Puig J, Patel S, Uddin A, Zhang J. Safety and efficacy of aliskiren/amlodipine/hydrochlorothiazide triple combination in patients with moderate to severe hypertension: a 54-week, open-label study. J Clin Hypertens (Greenwich). 2012 Dec;14(12):821-7. doi: 10.1111/j.1751-7176.2012.00706.x. Epub 2012 Aug 28. PMID 23205748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with essential hypertension were enrolled in the study at 82 investigative sites worldwide from 5 June 2008 to 5 October 2009.
Pre-assignment Details: A total of 635 participants entered the washout period, of which 564 participants met the study entry criteria and entered the study treatment phase.
Groups:
- Aliskiren /Amlodipine/Hydrochlorothiazide: Participants received aliskiren 300 milligrams (mg) plus hydrochlorothiazide 12.5 mg for one week, at Week 1 followed by combination of aliskiren 300 mg plus amlodipine 5 mg plus hydrochlorothiazide 12.5 mg for one week, at Week 2. Following Week 2, participants were force titrated up to aliskiren 300 mg plus amlodipine 10 mg plus hydrochlorothiazide 25 mg for 26 to 52 weeks (Weeks 28 to 54). All study medications were taken orally with water, once daily in the morning.
Period: Overall Study
Arm/Group | Aliskiren /Amlodipine/Hydrochlorothiazide
Started | 564
Completed | 493
Not Completed | 71
Not completed — Adverse Event | 39
Not completed — Abnormal Test Procedure | 1
Not completed — Unsatisfactory Therapeutic Effect | 3
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 17
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Population: Treated Population consisted of all participants who received at least one dose of trial medication.
Groups:
- Aliskiren /Amlodipine/Hydrochlorothiazide: Participants received aliskiren 300 mg plus hydrochlorothiazide 12.5 mg for one week, at Week 1 followed by combination of aliskiren 300 mg plus amlodipine 5 mg plus hydrochlorothiazide 12.5 mg for one week, at Week 2. Following Week 2, participants were force titrated up to aliskiren 300 mg plus amlodipine 10 mg plus hydrochlorothiazide 25 mg for 26 to 52 weeks (Weeks 28 to 54). All study medications were taken orally with water, once daily in the morning.
Arm/Group | Aliskiren /Amlodipine/Hydrochlorothiazide
Number analyzed (Participants) | 564
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238
  Male | 326

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs), Serious Adverse Events (SAEs) and Death
Description: An AE was defined as the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug, even if the event is not considered to be related to study drug. An SAE was defined as an event which was fatal or life-threatening, resulted in persistent or significant disability/incapacity, constituted a congenital anomaly/birth defect, required inpatient hospitalization or prolongation of existing hospitalization, was medically significant, i.e. defined as an event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: 54 weeks
Population: Treated Population consisted of all participants who received at least one dose of trial medication.
Measure: Count of Participants; unit: Participants
Groups:
- Aliskiren/Hydrochlorothiazide 300/12.5 mg: Participants received aliskiren 300 mg plus hydrochlorothiazide 12.5 mg, orally with water, once daily in the morning, for one week, at Week 1.
- Aliskiren/Amlodipine/Hydrochlorothiazide 300/5/12.5 mg: Following Week 1, participants received combination of aliskiren 300 mg plus amolodipine 5 mg plus hydrochlorothiazide 12.5 mg for one week, at Week 2. All study medications were taken orally with water, once daily in the morning.
- Aliskiren/Amlodipine/Hydrochlorothiazide 300/10/25 mg: Following Week 2, participants were force titrated up to aliskiren 300 mg plus amolodipine 10 mg plus hydrochlorothiazide 25 mg for 26 to 52 weeks (Weeks 28 to 54). All study medications were taken orally with water, once daily in the morning.
Arm/Group | Aliskiren/Hydrochlorothiazide 300/12.5 mg | Aliskiren/Amlodipine/Hydrochlorothiazide 300/5/12.5 mg | Aliskiren/Amlodipine/Hydrochlorothiazide 300/10/25 mg
Number analyzed (Participants) | 564 | 561 | 556
Participants
  Any Adverse Events | 57 | 54 | 255
  Serious Adverse Events | 0 | 1 | 14
  Death | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: The arm in which the highest sitting diastolic pressures were found at study entry was the arm used for all subsequent readings. A calibrated sphygmomanometer and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the participant in a sitting position for five minutes, systolic/diastolic blood pressure were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements. A negative change indicates improvement. Week 28 Endpoint was the last non-missing post-baseline measurement value on or before Week 28, and Week 54 Endpoint was the last non-missing measurement value after Week 28.
Time Frame: Baseline, Weeks 28 and 54 endpoint
Population: Treated Population consisted of all participants who received at least one dose of trial medication. Number analyzed is the number of participants with data available at both baseline and post-baseline time points.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Aliskiren/Amlodipine/Hydrochlorothiazide: Participants received aliskiren 300 mg plus hydrochlorothiazide 12.5 mg for one week, at Week 1 followed by combination of aliskiren 300 mg plus amlodipine 5 mg plus hydrochlorothiazide 12.5 mg for one week, at Week 2. Following Week 2, participants were force titrated up to aliskiren 300 mg plus amlodipine 10 mg plus hydrochlorothiazide 25 mg for 26 to 52 weeks (Weeks 28 to 54). All study medications were taken orally with water, once daily in the morning.
Arm/Group | Aliskiren/Amlodipine/Hydrochlorothiazide
Number analyzed (Participants) | 564
mmHg
  Baseline | 101.8 (7.74)
  Change from Baseline to Week 28 Endpoint | -20.3 (8.92)
  Change from Baseline to Week 54 Endpoint: number analyzed (Participants) | 205
  Change from Baseline to Week 54 Endpoint | -21.8 (8.66)

3. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 2
Time Frame: Baseline, Weeks 28 and 54 endpoints
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Aliskiren/Amlodipine/Hydrochlorothiazide
Number analyzed (Participants) | 564
millimeters of mercury
  Baseline | 166.1 (11.59)
  Change from baseline to Week 28 Endpoint | -34.2 (14.16)
  Change from Baseline to Week 54 Endpoint: number analyzed (Participants) | 205
  Change from Baseline to Week 54 Endpoint | -37.3 (14.63)

4. Secondary Outcome: Percentage of Participants Achieving the Blood Pressure Control Target of <140/90 mmHg
Description: Blood pressure control was defined as having a mean sitting diastolic blood pressure <90 mmHg and a mean sitting systolic blood pressure <140 mmHg. Percentage of participants achieving the blood pressure control of < 140/90 mmHg were reported. Week 28 Endpoint was the last non-missing post-baseline measurement value on or before Week 28 and Week 54 Endpoint was the last non-missing measurement value after Week 28.
Time Frame: Weeks 28 and 54 endpoints
Population: Treated Population consisted of all participants who received at least one dose of trial medication. Number analyzed is the number of participants with data available at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren/Amlodipine/Hydrochlorothiazide
Number analyzed (Participants) | 564
percentage of participants
  Week 28 Endpoint | 69.1
  Week 54 Endpoint: number analyzed (Participants) | 205
  Week 54 Endpoint | 77.1

5. Secondary Outcome: Percentage of Participants Who Achieved a Blood Pressure Response in Mean Sitting Diastolic Blood Pressure
Description: Diastolic Blood pressure response was defined as a mean sitting diastolic blood pressure <90 mmHg or a >=10 mmHg reduction from baseline value. Week 28 Endpoint was the last non-missing post-baseline measurement value on or before Week 28, and Week 54 Endpoint was the last non-missing measurement value after Week 28.
Time Frame: Weeks 28 and 54 endpoints
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren/Amlodipine/Hydrochlorothiazide
Number analyzed (Participants) | 564
percentage of participants
  Week 28 Endpoint | 91.8
  Week 54 Endpoint: number analyzed (Participants) | 205
  Week 54 Endpoint | 96.6

6. Secondary Outcome: Percentage of Participants Who Achieved a Blood Pressure Response in Mean Sitting Systolic Blood Pressure
Description: Systolic blood pressure response was defined as a mean sitting systolic blood pressure <140 mmHg or a >=20 mmHg reduction from baseline value. Week 28 Endpoint was the last non-missing post-baseline measurement value on or before Week 28, and Week 54 Endpoint was the last non-missing measurement value after Week 28.
Time Frame: Weeks 28 and 54 endpoints
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren/Amlodipine/Hydrochlorothiazide
Number analyzed (Participants) | 564
percentage of participants
  Week 28 Endpoint | 90.2
  Week 54 Endpoint: number analyzed (Participants) | 205
  Week 54 Endpoint | 93.7

ADVERSE EVENTS:
Time Frame: From Baseline up to 54 weeks.
Arm/Group | Aliskiren/Hydrochlorothiazide 300/12.5 mg | Aliskiren/Amlodipine/Hydrochlorothiazide 300/5/12.5 mg | Aliskiren/Amlodipine/Hydrochlorothiazide 300/10/25 mg
All-Cause Mortality (participants affected / at risk) | 0/564 | 0/561 | 0/556
Serious Adverse Events (participants affected / at risk) | 0/564 | 1/561 | 14/556
Other Adverse Events (participants affected / at risk) | 21/564 | 14/561 | 141/556
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Hydrochlorothiazide 300/12.5 mg (N=564) | Aliskiren/Amlodipine/Hydrochlorothiazide 300/5/12.5 mg (N=561) | Aliskiren/Amlodipine/Hydrochlorothiazide 300/10/25 mg (N=556)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 2
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Drug dependence (Psychiatric disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Hydrochlorothiazide 300/12.5 mg (N=564) | Aliskiren/Amlodipine/Hydrochlorothiazide 300/5/12.5 mg (N=561) | Aliskiren/Amlodipine/Hydrochlorothiazide 300/10/25 mg (N=556)
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 11
Oedema peripheral (General disorders) | 1 | 0 | 52
Bronchitis (Infections and infestations) | 2 | 3 | 16
Influenza (Infections and infestations) | 0 | 0 | 15
Nasopharyngitis (Infections and infestations) | 3 | 2 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 12
Headache (Nervous system disorders) | 10 | 6 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.